CLINICAL TRIAL: NCT05069012
Title: Optimal Dose of Intrathecal Morphine for Postoperative Analgesia After Cesarean Delivery
Brief Title: Intrathecal Morphine for Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Hess, Associate Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P000688
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Pain
Keywords: cesarean; morphine; multimodal analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Intervention Model Description: Prospective randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization maintained in the research pharmacy. Blinded syringe delivered to the investigator for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 50 micrograms (Active Comparator): Patients in this arm will receive 50 micrograms of morphine administered in the spinal fluid as part of their anesthesia for cesarean delivery
  Interventions: Drug: Morphine Sulfate
- 150 micrograms (Active Comparator): Patients in this arm will receive 150 micrograms of morphine administered in the spinal fluid as part of their anesthesia for cesarean delivery
  Interventions: Drug: Morphine Sulfate
- 250 micrograms (Active Comparator): Patients in this arm will receive 250 micrograms of morphine administered in the spinal fluid as part of their anesthesia for cesarean delivery
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Morphine Sulfate — Morphine is administered to provide pain relief after cesarean delivery; this is an assessment of the dose-response as measured by the duration of pain relief

SUMMARY:
This is a randomized double blinded non-inferiority study comparing the duration of pain relief when patients receive one of three doses of spinal morphine. Enrolled patients will be randomly assigned to receive either 50 mcg, 150 mcg, or 250 mcg. All patients will receive standardized postoperative care, including multimodal analgesia. The primary outcome will be the time until the patient requests additional opioid pain medications.

DETAILED DESCRIPTION:
Prospective, randomized, double-blind, controlled trial, with a non-inferiority design. Patients will be randomly assigned to receive either intrathecal morphine 50 mcg, 150 mcg, or 250 mcg based on a pre-assigned randomization sequence. This medication will be administered as part of their spinal anesthesia for cesarean delivery. the patient, clinician who administers the spinal anesthesia, and investigator who follows the patient will all be blinded to the dose of medication.

All patients will receive standard of care for cesarean delivery and routine nursing care. This includes: preoperative intravenous catheter placement with preoperative IV fluid, standard American Society of Anesthesiologists monitoring, and neuraxial anesthesia placement (either spinal or combined spinal epidural) in sterile fashion. Each patient will receive standard cesarean induction dose of intrathecal medication consisting of 1.5ml of 0.75% hyperbaric bupivacaine, fentanyl 25 mcg. At end of surgery, all patients will receive standard dose of ketorolac 30 mg IV and acetaminophen 1 gm IV and continue with redosing every 6 and 8 hours (respectively) for 24 hours. On arrival to PACU, all patients will receive standard nursing care with standard monitoring of side effects. On discharge from PACU, patients will be transferred to postpartum floor and receive standard nursing care and monitoring.

Over the following 24 hours, the patient will receive all standard post-cesarean care. For treatment of breakthrough pain, medications will provided be per standard care: oxycodone 5-10 mg PO every four hours PRN for pain. If the patient is not comfortable after receiving oral oxycodone they will be assessed by an anesthesia provider for either regional nerve block or additional opioids, as a one-time dose or by patient controlled analgesia (PCA).

For treatment for side effects, medications will provided be per standard care: ondansetron 4mg IV as first-line for nausea/vomiting, promethazine 6.25 mg IV or Haloperidol 0.5-1mg IV for refractory nausea/vomiting. Naloxone 0.04 mg IV for refractory pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women (ASA 2)
* Between 18 and 45 years old
* Singleton term pregnancies
* Planned neuraxial anesthesia

Exclusion Criteria:

* Refusal to participate
* Known allergy or contraindication to any medication used in the study
* Significant medical or obstetrical disease (ASA ≥ 3)
* Opioid use disorder
* Chronic pain syndrome
* Daily or near daily opioid use within last 3 weeks.
* Patient receiving a Monoamine oxidase inhibitors (MOAi)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-07-23 (Actual); Study Completion 2022-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borrelli MC, Sprowell AJ, Moldysz A, Idris M, Armstrong SL, Kowalczyk JJ, Li Y, Hess PE. A randomized controlled trial of spinal morphine with an enhanced recovery pathway and its effect on duration of analgesia after cesarean delivery. Anaesth Crit Care Pain Med. 2024 Feb;43(1):101309. doi: 10.1016/j.accpm.2023.101309. Epub 2023 Oct 18. PMID 37863195

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 50 Micrograms | 150 Micrograms | 250 Micrograms
Started | 24 | 24 | 24
Completed | 23 | 23 | 24
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Two patients were not analyzed due to pre-defined exclusion criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 Micrograms | 150 Micrograms | 250 Micrograms | Total
Number analyzed (Participants) | 23 | 23 | 24 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.0 (3.8) | 33.9 (4.8) | 36.8 (4.9) | 35.6 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 24 | 70
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 6
  Not Hispanic or Latino | 21 | 20 | 23 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 2 | 7
  White | 12 | 16 | 19 | 47
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 3 | 4 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Duration of Pain Relief
Description: Time to patient request for first dose of oral rescue pain medicine
Time Frame: 72 hours after delivery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | 50 Micrograms | 150 Micrograms | 250 Micrograms
Number analyzed (Participants) | 23 | 23 | 24
hours | 24.5 [3.5 to 34.4] | 29.4 [24.5 to 72] | 32 [30.5 to 72]

2. Secondary Outcome: Pain Scores
Description: Visual analogue pain scores reported by the patient. Scale measured on a line from 0 to 100 mm, with 0 representing 'no pain' and 100 representing 'worst possible pain'
Time Frame: 24 hours after delivery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms | 150 Micrograms | 250 Micrograms
Number analyzed (Participants) | 23 | 23 | 24
score on a scale | 2.2 [1.3 to 5.1] | 1.8 [0.8 to 2.3] | 1.9 [0.2 to 2.9]

3. Secondary Outcome: Quality of Recovery
Description: Quality of Recovery Score following Cesarean Delivery Questionnaire (ObsQoR-11). This is a multi-dimensional wellness scale ranging from 0 (worst) to 120 (best) along 12 axis items.
Time Frame: 24 hours after delivery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms | 150 Micrograms | 250 Micrograms
Number analyzed (Participants) | 23 | 23 | 24
score on a scale | 72 [38 to 87] | 93 [83 to 109] | 95 [85 to 102]

4. Secondary Outcome: Nausea
Description: Incidence of nausea and vomiting requiring treatment with a medication
Time Frame: 24 hours after delivery
Measure: Number; unit: percentage of participants
Arm/Group | 50 Micrograms | 150 Micrograms | 250 Micrograms
Number analyzed (Participants) | 23 | 23 | 24
percentage of participants | 4.3 | 8.7 | 12.5

5. Secondary Outcome: Pruritus
Description: Incidence of pruritus requiring treatment with a medication
Time Frame: 24 hours after delivery
Measure: Number; unit: percentage of participants
Arm/Group | 50 Micrograms | 150 Micrograms | 250 Micrograms
Number analyzed (Participants) | 23 | 23 | 24
percentage of participants | 8.7 | 4.3 | 4.1

ADVERSE EVENTS:
Time Frame: 24 hours after delivery
Arm/Group | 50 Micrograms | 150 Micrograms | 250 Micrograms
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT05069012/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT05069012/ICF_001.pdf